CLINICAL TRIAL: NCT03394378
Title: The Impact of Non-Alcoholic Fatty Pancreas Disease on Outcome of Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ningbo3
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Non-Alcoholic Fatty Pancreas Disease; Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Obesity is a well-established risk factor for acute pancreatitis (AP). As for non-alcoholic fatty pancreas disease (NAFPD), it is evident that it is correlated with obesity. This is apparently the first study evaluating the association between NAFPD and severity of AP after taking into account several covariates.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a common disease with a highly variable clinical course, which can range from a mild, self-limited disease to severe disease with a mortality rate of 10-20%. It is vital to distinguish severe cases early because they require more aggressive fluid resuscitation and early nutritional support.

Obesity is a well-established risk factor for acute pancreatitis (AP). It leads to ectopic fat accumulation in visceral organs, such as the liver, skeletal muscles, heart and pancreas.

Assuming that attenuation in the pancreas seen on unenhanced computed tomography (CT) scanning is inversely associated with severe outcomes in AP, we investigated the relationship between NAFPD and severity of AP and the significance of pancreas attenuation for the prognosis and mortality in AP patients. The result of this study suggest that decreased pancreas attenuation and P/S ratio are strong predictors of severe pancreatitis, mortality, systemic complication.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with AP
2. age>18y

Exclusion Criteria:

1. age<18y
2. missing data in the electronic medical record
3. prior attacks of AP
4. without spleen
5. with ambiguous pancreatic margin

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosis criteria for AP were the presence of at least 2 of the 3 following factors: (1) abdominal pain characteristic of AP, (2) serum amylase and/or lipase levels>= 3 times the upper limit of normal, and (3) characteristic findings of AP on a CT scan
Sampling Method: Non-Probability Sample
Enrollment: 1662 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Comparison of characteristics and variables according to severity of AP. | the physical examination data in the year of 2017
  Comparison of characteristics and variables according to severity of AP by One-Way Analysis of variance(ANOVA) and Pearson chi-square test.
The association between pancreas attenuation and ICU transfer, pancreatitis severity, systemic and local complications and prognostic scores (APACHE II scores, Ranson score, BISAP score and SIRS). | the physical examination data in the year of 2017
  The association between pancreas attenuation and ICU transfer, pancreatitis severity, systemic and local complications and prognostic scores (APACHE II scores, Ranson score, BISAP score and SIRS) by Likelihood Ratio test.
BMI adjusted hazard ratios (HRs) and 95% CIs for the relationship between NAFPD and mortality of acute pancreatitis, evaluated by pancreas attenuation (HU), P/S ratio. | the physical examination data in the year of 2017
  BMI adjusted hazard ratios (HRs) and 95% CIs for the relationship between NAFPD and mortality of acute pancreatitis, evaluated by pancreas attenuation (HU), P/S ratio by cox proportional hazards models.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xu, Dr, Principal Investigator — Department of gastroenterology,Ningbo No.1 Hospital, Ningbo, China
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China